CLINICAL TRIAL: NCT03791268
Title: The Establishment of General Tissue Response Classification System After Chemotherapy According to Gastric Cancer Patients With Neoadjuvant Chemotherapy
Brief Title: General Tissue Response Classification System After Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jian-Kun Hu, Vice director of Gastrointestinal Surgery department, West China Hospital; Director of Institute of Gastric Cancer, State Key Laboratory of Biotherapy, West China Hospital, West China Hospital
Other Study IDs: WCH-GC-06
Record Dates: First submitted 2018-12-25; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Stomach Adenocarcinoma
Keywords: Stomach Adenocarcinoma; neoadjuvant chemotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Gastric Cancer Patients who underwent Chemotherapy and will have gastric cancer surgery.
  Interventions: Procedure: Gastric cancer surgery

INTERVENTIONS:
Procedure: Gastric cancer surgery — Gastric cancer surgery is performed according to the Japanese Guidelines. Patients will intraoperative evaluate the edema, fibrosis and exudation.

SUMMARY:
This research intend to collect the information of gastric cancer patients who received preoperative neoadjuvant chemotherapy and radical gastric ectomy at Department of Gastrointestinal Surgery, West China Hospital, Sichuan University. Base on The degree of edema, intraoperative effusion, fibrosis of connecting tissues, the investigators aim to constitute the core parameters of the tissue response grading system following neoadjuvant chemotherapy, and explore the mutual effect among the tissue response grading system, tumor regression response and long-term survival outcome of tumor patients.

DETAILED DESCRIPTION:
Gastric cancer is ranked the third malignancy carcinoma which related deaths. In china, gastric cancer always ranked in the top three cancer-related deaths. Early diagnosis ratio of gastric caner is low in china. And the proportion of gastric cancer cases which performed surgical treatment is less than 20% at early stage Therefore, the vast majority of patients with gastric carcinoma already have locally advanced tumors at the time of diagnosis in china, and the current treatment strategy is suggested to receive comprehensive surgical gastrectomy. Current research showed strong evidence that preoperative neoadjuvant therapy represented by neoadjuvant chemotherapy (NAC) can downstaging the primary tumor to increase the possibility of a successful complete resection and destroying occult lymph node and distant micro metastases to decrease the rate of tumor recurrence., and thus provide the survival benefit for locally advanced gastric cancer patients.Therefore, the national comprehensive cancer network(NCCN)guidelines for gastric cancer treatment(2017 version 5),recommended that neoadjuvant chemotherapy (evidential level category 1 ) and neoadjuvant chemotherapy (evidential level category 2B) can be considered.for locally advanced gastric caner cases(T2-4nx).

Through the literature review, the investigators found that residual tumor evaluation criteria which was promoted by Becker and the criteria for tumor regression response which recommended by NCCN guidelines can be used to evaluate the tumor regression after chemotherapy/radiotherapy. However, the rating criteria for connective tissue response around the tumor after chemotherapy/radiotherapy still remain blank area. During the clinical practice, surgeons should not ignored the edema and fibrosis of tumor and connective tissue after chemotherapy/radiotherapy which existed objectively. Recent research generally believed that preoperative chemotherapy with/or not with radiotherapy may lead to edema of gastrointestinal tract and perigastric tissues, intraoperative effusion and fibrosis of tumor and lymph nodes bearing tissues，which may increase the difficulty of tissue dissociation and lymph node dissection, increase the risk of surgical trauma, and may lead to increased incidence of postoperative complications. There is till a lack of evaluation criteria for the degree of tissue fibrosis/edema after radiotherapy and chemotherapy which may have impact on surgery and long-term survival prognosis of patients.

Therefore, it is necessary to analyze and evaluate tissue edema and fibrosis after chemotherapy/radiotherapy and establish corresponding criteria system to explore whether if the tissue fibrosis and edema are involved with the degree of tumor retreat after chemotherapy/radiotherapy at two aspects: general evaluation and histopathology. The interaction effects of tissue fibrosis and edema with the difficulty of operation and incidence rate of postoperative complications. In addition, the mutual effect of tissue fibrosis and edema with the final long-term survival outcome of tumor patients needs to be evaluated from two aspects: general observation and histopathology evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of gastric cancer was clear，Patients with definitely clinical evidence of locally advanced disease (cT3 ⁄ 4、N-/+、M0).
2. Preoperative chemotherapy has been administered，and intended to receive surgical resection.
3. Age:less than or equal to 75 years old and more than 18 years old;
4. Without any other malignant tumor, without any serious concomitant disease.
5. Eastern Cooperative Oncology Group (ECOG) physical status score <2, America Society of Anesthesiologist (ASA) score<3
6. No restriction on gender or race; Informed consent has been signed by patient or entrusted agent；

Exclusion Criteria:

1. Previous history of gastric ulcer or gastric perforation;
2. Previous operation history at upper abdominal, except laparoscopic cholecystectomy;
3. Emergency operation caused by obstruction, perforation,and acute hemorrhage;
4. The patient can not tolerate the surgical treatment which caused by other serious concomitant disease, such as severe pulmonary disease, cardiac clinical function below are below level 2, pulmonary infection, moderate or severe chronic obstructive pulmonary disease (COPD), chronic bronchitis
5. Patient has severe mental illness
6. The patient and agent request to withdraw from the clinical study after signing the consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients who received preoperative neoadjuvant chemotherapy and radical gastric ectomy at Department of Gastrointestinal Surgery, West China Hospital, Sichuan University
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
General observation of tissue fibrosis, edema and exudation (Intraoperation) | The 1 day of surgery
  To assess the degree of fibrosis, edema and exudation in tumor tissue and main perigastric lymph node area during the operation.

SECONDARY OUTCOMES:
General observation of tissue edema (Intraoperation) | The 1 day of surgery
  To assess the degree of edema in tumor tissue and main perigastric lymph node area during the operation.
General observation of tissue exudation (Intraoperation) | The 1 day of surgery
  To assess the degree of exudation in tumor tissue and main perigastric lymph node area during the operation.
Histopathology evaluation of edema | The 1 day of surgery
  To assess the degree of edema in tumor tissue and main perigastric lymph node area by pathological section.
Histopathology evaluation of tissue fibrosis | Postoperative 30 days
  To assess the degree of fibrosis in tumor tissue and main perigastric lymph node area by pathological section.
Postoperative mortality rate | Postoperative 30 days
  Calculated by the number of patients with any operative complication as the numerator and the number of patients undergoing surgical treatment.
Survival outcome | Postoperative 3 Years
  The 3-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang H, Zhang WH, Ge R, Peng BQ, Chen XZ, Yang K, Liu K, Chen XL, He D, Liu JP, Zhang WW, Qin Y, Zhou ZG, Hu JK. Application of Gross Tissue Response System in Gastric Cancer After Neoadjuvant Chemotherapy: A Primary Report of a Prospective Cohort Study. Front Oncol. 2021 Nov 24;11:585006. doi: 10.3389/fonc.2021.585006. eCollection 2021. PMID 34900661